CLINICAL TRIAL: NCT00773773
Title: A Study to Assess if a Combination of Serum Measurements of Molecular Biomarkers and Serum Protein Profiling Can be Used to Predict Which Patients Undergoing Prostatic Biopsy Will be Diagnosed With Cancer
Brief Title: Combination of Serum Measurements of Molecular Biomarkers and Serum Protein Profiling Can be Used to Predict Which Patients Undergoing Prostatic Biopsy Will be Diagnosed With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol closed to accrual early due to PI retirement.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other); State University of New York - Downstate Medical Center (Other); NYU Langone Health (Other); Kings County Hospital Department of Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-114
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Elevated Prostate Specific Antigen (PSA)
Keywords: Biomarkers - PSA, hK2 and solubilized; urokinase-receptor forms (su-PAR); 08-114
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Patients undergoing prostatic biopsy (Experimental): This study will enroll two groups of 250 patients who are to undergo prostatic biopsy as part of their routine medical care because of suspicion of prostate cancer (elevated PSA between 2 and 10 ng/ml, abnormal rectal examination, or both). The first group will contain 250 patients of African-American descent and the second will contain 250 Caucasian men.
  Interventions: Other: serum specimens obtained will be utilized for proteomic profiling comprising MALDI-TOF MS, and serum biomarker assays.

INTERVENTIONS:
Other: serum specimens obtained will be utilized for proteomic profiling comprising MALDI-TOF MS, and serum biomarker assays. — Patients referred for prostate biopsy as part of their routine care are to be recruited. Patients will undergo standard medical evaluation/care by undergoing a prostate biopsy because of an elevated PSA blood test and/or an abnormal digital rectal prostate examination. The protocol involves obtaining the research blood sample at the time of routine pre-biopsy blood draw. As such, an extra five (40 mL) tubes of blood will be drawn. The serum specimens obtained will be utilized for proteomic profiling comprising MALDI-TOF MS, and serum biomarker assays.

SUMMARY:
This is a prospective, serum proteomics study of men who are to undergo prostate biopsy. The purpose is to determine if proteomic profiles can be used to distinguish between men with prostate cancer on biopsy from men with no cancer on biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older
* Have a PSA level between 2 and 10 ng/ml
* May or may not have an abnormal digital rectal examination
* Scheduled for trans-rectal ultrasound (TRUS) guided systematic prostate biopsy as part of routine medical care. All sites (Department of Urology at SUNY Downstate Medical Center, Brooklyn, the Department of Urology, New York Presbyterian Hospital, Weill Medical College of Cornell University, Manhattan and the Department of Urology, Kings County Hospital) will perform a standardized 14 core biopsy protocol.
* Signed, informed consent
* Patient must be able to attend the pre-biopsy blood draw

Exclusion Criteria:

* Any period of prior/current treatment with hormonal therapy (LHRH agonist/antagonist,antiandrogen, 5-alpha-reductase inhibitor)
* Prior pelvic radiation
* A period of less than 6 months prior/current treatment with an alpha-blocker
* Previous diagnosis of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-10-14 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tempst, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Kings County Hopsital Center, Brooklyn, New York
  - SUNY Downstate Medical Center (DMC), Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Weill Medical College of Cornell University, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Undergoing Prostatic Biopsy
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 65 [49 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 54
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Men With Prostate Cancer Have a Different Proteomic Profile Than Men Without Cancer. Cancer-free Status Will be Confirmed by a Re-biopsy at 6 Months to Reduce the Biopsy False Negative Rate to Less Than 5 %.
Time Frame: conclusion of study
Population: N/A - data were not collected
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 0

2. Primary Outcome: To Determine Whether the Peptide Proteomic Profile Can Improve the Predictive Ability of Known Serum Biomarkers (PSA (Free and Total), hK2 and Su-PAR) for Prostate Cancer.
Time Frame: conclusion of the study
Population: N/A - data were not collected
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 0

3. Secondary Outcome: To Determine if Caucasian Men and Men of African-American Descent With and Without Prostate Cancer Have Different Proteomic Profiles.
Time Frame: conclusion of the study
Population: N/A - data were not collected
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 0

4. Secondary Outcome: To Assess Reproducibility of Proteomic Profiles Over Different Runs, Platforms, and Sites.
Time Frame: conclusion of the study
Population: N/A - data were not collected
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 0

5. Secondary Outcome: To Procure a DNA Repository From These Patients Undergoing Prostate Biopsy for Future Assessment of Kallikrein Gene Expression.
Time Frame: conclusion of the study
Population: N/A - data were not collected
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 0

6. Secondary Outcome: To Establish a Bank of DNA, Serum, and Frozen Lymphoblastoid Cells From These Patients for the Purpose of Enabling Genetic Investigations in Men With a Diagnosis of Prostate Cancer.
Time Frame: conclusion of the study
Population: N/A - data were not collected
Arm/Group | Patients Undergoing Prostatic Biopsy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 years
Arm/Group | Patients Undergoing Prostatic Biopsy
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT00773773/Prot_SAP_000.pdf